CLINICAL TRIAL: NCT05811871
Title: Examining Variables Affecting Patient Participation in Clinical Trials for Tinnitus
Brief Title: Assessing Factors in Tinnitus Patients' Clinical Study Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84411336
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Tinnitus
Keywords: tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials can sometimes favor certain demographic groups. Additionally, there is limited research that delves into the factors that influence participation in clinical trials, both positive and negative.

The goal is to identify the obstacles and challenges that prevent participation in tinnitus clinical studies, as well as the reasons for withdrawal or discontinuation.

The insights gained from this study will ultimately benefit those with tinnitus who may be invited to participate in clinical research in the years to come.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with tinnitus
* Willing to comply with all study related procedures and assessments
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* No documented diagnosis of tinnitus
* Any other health problems that would prohibit safe participation in the study
* Pregnant or planning to become pregnant while enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tinnitus patients who are actively considering participating in an observational medical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of tinnitus patients who decide to enroll in a clinical study | 3 months
Rate of tinnitus patients who remain in a clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Natalini E, Fioretti A, Riedl D, Moschen R, Eibenstein A. Tinnitus and Metacognitive Beliefs-Results of a Cross-Sectional Observational Study. Brain Sci. 2020 Dec 23;11(1):3. doi: 10.3390/brainsci11010003. PMID 33374519
- [Background] Farr MR, Moraleda Deleito J, Xu Y, Ray J. Developing a one-stop tinnitus service: outcomes of a joined up management strategy: a retrospective observational cohort study. J Eval Clin Pract. 2016 Feb;22(1):93-97. doi: 10.1111/jep.12442. Epub 2015 Aug 28. PMID 26314274
- [Background] Tinnitus Retraining Therapy Trial Research Group; Scherer RW, Formby C. Effect of Tinnitus Retraining Therapy vs Standard of Care on Tinnitus-Related Quality of Life: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2019 Jul 1;145(7):597-608. doi: 10.1001/jamaoto.2019.0821. PMID 31120533

DOCUMENTS (1):
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT05811871/ICF_000.pdf